CLINICAL TRIAL: NCT01681524
Title: A Phase 3, Open Label, Multicenter Study for the Assessment of Myocardial Perfusion Using Positron Emission Tomography (PET) Imaging of Flurpiridaz F18 Injection in Patients With Suspected or Known Coronary Artery Disease (CAD)
Brief Title: Open Label Study to Access Flurpiridaz F18 in PET MPI Verses SPECT MPI
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: delayed study start
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BMS747158-302
Record Dates: First submitted 2012-08-28; First posted 2012-09-10 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease
Keywords: Flurpiridaz F18 Injection; Positron Emission Tomography Myocardial Perfusion Imaging; Single Positron Emission Computed Tomography; Coronary Artery Disease; Myocardia Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases | interventions — BMS 747158-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flurpiridaz F18 (Experimental): Open-label study of a single injection of flurpiridaz F18 for PET MPI compared to SPECT MPI in patients with suspected or known coronary artery disease referred for coronary cathertization
  Interventions: Drug: Flurpiridaz F18

INTERVENTIONS:
Drug: Flurpiridaz F18 — Injection of Flurpiridaz F18 for the purposes of PET MPI analysis

SUMMARY:
The study will evaluate the use of Flurpiridaz F18 injection in patients with CAD to determine if the study drug in PET imaging is better than SPECT imaging currently used for this purpose.

DETAILED DESCRIPTION:
The study will assess the diagnostic efficacy (sensitivity and specificity) of Flurpiridaz F18 Injection MPI in comparison with SPECT MPI in patients with known or suspected CAD. Six hundred and seventy-two evaluable patients will be enrolled and will undergo SPECT MPI and Flurpiridaz F18 PET MPI. Patients will be considered for enrollment if they are scheduled to undergo or have undergone prior ICA without intervention (being either positive or negative for CAD).

ELIGIBILITY:
Inclusion Criteria:

Invasive Coronary Angiography Men or Women age 18 or older - see protocol for additional details

Exclusion Criteria:

Women who are pregnant, lactating, or of child bearing potential who are not practicing birth control Unstable cardiac status History of coronary artery bypass graft History of PCI within the past six months See protocol for additional details

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Blinded Image assessment for PET & SPECT perfusion and for interventional coronary angiography | 12 months

SECONDARY OUTCOMES:
Diagnostic performance evaluation of CAD (PETVsSPECT) | 12 months
Diagnositic performance evaluation of multivessel disease (PETvsSPECT) | 12 months
Detection of CAD in subgroups: pharm stress, females and BMI>/=30 | 12 months
Image quality of rest and stress (PETvsSPECT) | 12 months
Diagnostic certainty evaluation of rest and stress (PETvsSPECT) | 12 months
Evaluation of reversible defect size of rest and stress (PETvsSPECT) | 12 months
Safety evaluation of flurpiridaz F 18 will include monitoring the number participants with adverse events (AEs), medication errors, treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Orlandi, MD, Study Director — Lantheus Medical Imaging